CLINICAL TRIAL: NCT03814642
Title: A Randomized, Open-label, Three-period, Multiple Dosing Crossover Clinical Trial to Evaluate the Influence of Tegoprazan on the Pharmacodynamics of Clopidogrel According to CYP2C19 Genotypes in Healthy Male Volunteers
Brief Title: Effect of Tegoprazan on Pharmacodynamics of Clopidogrel in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_110
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel; tegoprazan; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clopidogrel 75 mg (Active Comparator): Oral administration of clopidogrel 75 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg
- Clopidogrel 75 mg + Tegoprazan 50 mg (Experimental): Oral administration of clopidogrel 75 mg tablet and tegoprazan 50 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg; Drug: Tegoprazan 50 mg
- Clopidogrel 75 mg + Esomeprazole 20 mg (Experimental): Oral administration of clopidogrel 75 mg tablet and esomeprazole 20 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75 mg; Drug: Esomeprazole 20 mg

INTERVENTIONS:
Drug: Clopidogrel 75 mg — Clopidogrel 75 mg tablet
  Other Names: Plavix
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Clopidogrel 75 mg + Tegoprazan 50 mg
Drug: Esomeprazole 20 mg — Esomeprazole 20 mg tablet
  Other Names: Nexium
  Arms: Clopidogrel 75 mg + Esomeprazole 20 mg

SUMMARY:
This study aims to evaluate the influence of tegoprazan on the pharmacodynamics of clopidogrel according to CYP2C19 genotypes following co-administration of tegoprazan and clopidogrel in healthy male volunteers.

DETAILED DESCRIPTION:
Evaluation Criteria:

* Pharmacodynamic assessments using P2Y12 assay
* Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged ≥ 19 years and ≤ 50 years on the date of the written informed consent
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2 at the time of screening
* Helicobacter pylori negative
* Voluntarily decided to participate in the study and provided written informed consent before any screening procedure
* Judged by the investigator to be eligible for this study based on physical examination, laboratory test, inquiry, etc.

Exclusion Criteria:

* Has a history of or currently has clinically significant liver, kidney, nervous system, respiratory system, endocrine system, blood, cardiovascular system, urinary system, or psychiatric disease or tumor
* Has a history of or currently has gastrointestinal disorder (gastrointestinal ulcer, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.) that may influence the safety and pharmacodynamic assessments of the investigational product
* Has a history of gastrointestinal surgery (except simple appendectomy and hernia surgery)
* Hypersensitivity to drugs including the ingredients of the investigational product and other drugs (aspirin, antibiotics, etc.) or a history of clinically significant hypersensitivity
* Positive serological test including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Blood total bilirubin, AST (GOT), and ALT (GPT) levels greater than 1.5x of the upper limit of normal range at screening
* Platelet, PT and aPTT levels outside the upper/lower limit of normal range by 10% at screening
* P2Y12 Reaction Unit (PRU) by P2Y12 assay outside the upper/lower limit of normal range by 10% at screening
* *17 allele by CYP2C19 genotyping (Ultrarapid metabolizer)
* Systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 95 mmHg, or pulse rate < 45 beats/minute or > 100 beats/minute when vital signs are measured in sitting position after resting for at least 5 minutes during screening
* QTc > 450 msec, PR interval > 200 msec, QRS interval > 120 msec, and other clinically significant findings on electrocardiogram at screening
* Has a history of or positive urine screening for drug abuse
* Administration of any prescription drugs or herbal medicine within 2 weeks prior to the expected date of the first dose, or administration of any over-the-counter (OTC) drug, health functional food or vitamin within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise decided eligible by the investigator)
* Participation in other clinical study or bioequivalence study to receive an investigational product within 3 months prior to the expected date of the first dose
* Donation of whole blood within 2 months or apheresis/receipt of blood transfusion within 1 month prior to the expected date of the first dose
* Excessive caffeine intake (> 5 units/day) or persistent alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking during hospitalization period
* Smoking for more than 3 months prior to the study or inability to cease smoking throughout the study
* Inability to refrain from grapefruit-containing food from 24 hours before admission to discharge
* Inability to refrain from caffeine-containing food (coffee, tea (black tea, green tea, etc.), carbonated drink, coffee-flavored milk, nutritional tonic, etc.) from 24 hours before admission to discharge
* Inability to use a medically acceptable method of contraception throughout the study. Medically acceptable methods of contraception include use of intrauterine device with established failure rate of contraception by spouse (or partner), concomitant use of barrier method (for male or for female) and spermicide, or surgical procedure on subject himself or his partner (vasectomy, tubal resection/ligation, hysterectomy)
* Considered ineligible to participate in the study by the investigator based on laboratory test results or other reasons

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Change in P2Y12 Reaction Unit (PRU) from baseline | Pre-dose(0h) on days 1, 3, 5, and 8 in each period
  Pharmacodynamic blood sampling to measure PRU using VerifyNow® system

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea